CLINICAL TRIAL: NCT00531440
Title: A 2 Year Extension to a 1 Year Multicenter, Randomized, Open Label, Parallel Group Study of the Safety, Tolerability and Efficacy of Two Doses (1.5 and 3 mg/Day) of Everolimus (RAD001) With Basiliximab, Corticosteroids and Optimized Administration of Cyclosporine in de Novo Renal Transplant Recipients.
Brief Title: This is a 2-year Follow-up Study to Evaluate the Long-term Effects in Patients Who Completed the Study CRAD001A2307.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001A2307E1
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, everolimus, Immunosuppressants
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus (RAD001)

SUMMARY:
This extension study is designed to provide long-term safety and efficacy data beyond 12 months up to Month 36.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving study medication at Month 12 (CRAD001A2307) and sign a new Informed Consent to extend the treatment or observation period beyond Month 12.
* Female patients must agree to continue using an approved method of birth control throughout the study and for 3 months following the last dose of study medication.
* Another Informed Consent was required for the extension amendment. This Informed Consent allowed for separate consent to the amendment study itself, and the retrospective collection of biopsies and/or the yearly protocol biopsies.
* Inclusion and exclusion criteria were not changed, except that patients who completed the core study in follow-up became eligible to participate in the amended extension.

Exclusion Criteria:

* Patients who are receiving study medication and do not sign a new Informed Consent to extend the treatment and observation period beyond Month 12 cannot enter the extension.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2001-11; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
graft loss, death, biopsy-proven acute rejection,antibody-treated ,biopsy-proven chronic allograft nephropathy,retransplantation/dialysis up to 36m renal function measured by creatinine clearance Cockcroft-Gault)calculated glomerularfiltration rate

SECONDARY OUTCOMES:
biopsy-proven acute rejection episodes,graft loss, deathor lost to follow-up 6,12,24&3677 Mths both groups.assess the incidence of graft loss, death, biopsy-proven acute rejection, antibody-treated acute rejection, clinically-confirmed acute rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland